CLINICAL TRIAL: NCT03541772
Title: "Combined Oncoxin-Viusid® Treatment With Radiotherapy and Chemotherapy in Patients With Head and Neck Cancer. Phase II, Randomized and Double-blind Study"
Brief Title: Evaluation of Oncoxin-Viusid® in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-1
Record Dates: First submitted 2018-04-24; First posted 2018-05-31 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Head Cancer Neck
Keywords: Head Carcinoma; Neck Carcinoma; Chemotherapy; Radiotherapy; Oncoxin Viusid; Nutritional supplement
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncoxin-Viusid® (Experimental): Radiotherapy + Chemotherapy + Oncoxin-viusid®
  Interventions: Dietary Supplement: Oncoxin-Viusid®
- Placebo (Placebo Comparator): Radiotherapy + Chemotherapy + Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oncoxin-Viusid® — Radiotherapy for 6-8 weeks, chemotherapy for 1-22-43 days during Radiotherapy and Oncoxin-Viusid® (75 ml/day) before/during/after both treatments
  Arms: Oncoxin-Viusid®
Dietary Supplement: Placebo — Radiotherapy for 6-8 weeks, chemotherapy for 1-22-43 days during Radiotherapy and placebo (75ml/day) before/during/after both treatments
  Arms: Placebo

SUMMARY:
Nutritional supplements containing antioxidants seem to decrease toxicity associated with Radiotherapy (RT) and Chemotherapy (CT) in patients with malignant head and neck tumors. Oncoxin-Viusid® (OV) is a nutritional supplement with antioxidant, immunomodulator and antitumor effects.

DETAILED DESCRIPTION:
Objective

To assess the efficacy and safety of OV in patients with head and neck tumors during treatment with radio-chemotherapy.

Materials and Methods

Patients diagnosed with Head and Neck Carcinoma, and indicated to follow a radiotherapy treatment concurrent with Radiosensitizing Chemotherapy, were included in a phase II, randomized, prospective, controlled and double-blind study in two treatment arms: RT + CT + Placebo (n = 30) and RT + CT + OV (n = 30) during one year in a tertiary center (INOR), with the aim of evaluating the reduction of toxicities of RT-CT and improve the quality of life of patients during these oncospecific treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* over 18 years of age
* With histological diagnosis of carcinoma of the head and neck
* Regardless of the variety or degree of histological differentiation and clinical stage
* Tributaries of concomitant treatment with ionizing radiation and radiosensitizing chemotherapy with intercurrent diseases compensated and index of Karnofsky > 59
* Acceptable hematological parameters
* Women not pregnant or lactating
* Who authorized their inclusion in the investigation, through their informed consent.

Exclusion Criteria:

* Patients with a second concomitant primary tumor and / or contraindication to platinum chemotherapy
* Patients who are under another research protocol or who have decompensated psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Decrease the degrees of toxicities of Radiotherapy and Chemotherapy | 4 months
  Tumor biopsy
Decrease the degrees of toxicities of Radiotherapy and Chemotherapy | 4 months
  Biochemical analysis of urine
Decrease the degrees of toxicities of Radiotherapy and Chemotherapy | 4 months
  anamnesis
Decrease the degrees of toxicities of Radiotherapy and Chemotherapy | 4 months
  physical examination
Improve the quality of life of patients during radiotherapy | 4 months
  Index of Karnofsky

SECONDARY OUTCOMES:
Duration of the therapeutic range of radiotherapy | 4 months
  Kaplan-Meyer's Method

CONTACTS AND LOCATIONS:
Overall Officials: Ivonne Chon, Dr., Principal Investigator — INOR
Locations (1):
- National Institute of Oncology and Radiobiology of Cuba, Vedado, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Marin Caro MM, Laviano A, Pichard C. Nutritional intervention and quality of life in adult oncology patients. Clin Nutr. 2007 Jun;26(3):289-301. doi: 10.1016/j.clnu.2007.01.005. Epub 2007 Mar 21. PMID 17368656
- [Background] Brizel DM, Wasserman TH, Henke M, Strnad V, Rudat V, Monnier A, Eschwege F, Zhang J, Russell L, Oster W, Sauer R. Phase III randomized trial of amifostine as a radioprotector in head and neck cancer. J Clin Oncol. 2000 Oct 1;18(19):3339-45. doi: 10.1200/JCO.2000.18.19.3339. PMID 11013273
- [Background] Antonadou D, Pepelassi M, Synodinou M, Puglisi M, Throuvalas N. Prophylactic use of amifostine to prevent radiochemotherapy-induced mucositis and xerostomia in head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):739-47. doi: 10.1016/s0360-3016(01)02683-9. PMID 11849797
- [Background] Bardia A, Tleyjeh IM, Cerhan JR, Sood AK, Limburg PJ, Erwin PJ, Montori VM. Efficacy of antioxidant supplementation in reducing primary cancer incidence and mortality: systematic review and meta-analysis. Mayo Clin Proc. 2008 Jan;83(1):23-34. doi: 10.4065/83.1.23. PMID 18173999
- [Background] Lamson DW, Brignall MS. Natural agents in the prevention of cancer, part two: preclinical data and chemoprevention for common cancers. Altern Med Rev. 2001 Apr;6(2):167-87. PMID 11302780
- [Background] Marquez J, Mena J, Hernandez-Unzueta I, Benedicto A, Sanz E, Arteta B, Olaso E. Ocoxin(R) oral solution slows down tumor growth in an experimental model of colorectal cancer metastasis to the liver in Balb/c mice. Oncol Rep. 2016 Mar;35(3):1265-72. doi: 10.3892/or.2015.4486. Epub 2015 Dec 16. PMID 26676882
- [Background] Rodrigues MJ, Bouyon A, Alexandre J. [Role of antioxidant complements and supplements in oncology in addition to an equilibrate regimen: a systematic review]. Bull Cancer. 2009 Jun;96(6):677-84. doi: 10.1684/bdc.2009.0886. French. PMID 19493854
- [Background] Lamson DW, Brignall MS. Antioxidants in cancer therapy; their actions and interactions with oncologic therapies. Altern Med Rev. 1999 Oct;4(5):304-29. PMID 10559547
- [Background] Lamson DW, Brignall MS. Antioxidants and cancer therapy II: quick reference guide. Altern Med Rev. 2000 Apr;5(2):152-63. PMID 10767670
- [Background] Mahdavi R, Faramarzi E, Seyedrezazadeh E, Mohammad-Zadeh M, Pourmoghaddam M. Evaluation of oxidative stress, antioxidant status and serum vitamin C levels in cancer patients. Biol Trace Elem Res. 2009 Jul;130(1):1-6. doi: 10.1007/s12011-008-8309-2. Epub 2009 Jan 17. PMID 19148586
- [Background] Hernandez-Unzueta I, Benedicto A, Olaso E, Sanz E, Viera C, Arteta B, Marquez J. Ocoxin oral solution(R) as a complement to irinotecan chemotherapy in the metastatic progression of colorectal cancer to the liver. Oncol Lett. 2017 Jun;13(6):4002-4012. doi: 10.3892/ol.2017.6016. Epub 2017 Apr 10. PMID 28599406